CLINICAL TRIAL: NCT02461303
Title: Non-Invasive Methods to Maximize Fertility in Peri-Pubertal Patients With Klinefelter Syndrome
Brief Title: Fertility Assessment in Patients With Klinefelter Syndrome
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit the anticipated number of subjects for this study
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kyle Orwig, Professor, University of Pittsburgh
Other Study IDs: PRO15030141
Record Dates: First submitted 2015-05-26; First posted 2015-06-03 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Klinefelter Syndrome
Keywords: Klinefelter; Spermatogenesis; Puberty; Fertility
MeSH Terms: conditions — Klinefelter Syndrome | interventions — Counseling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Semen samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Counseling — Subjects will be counseled on the impact of KS on the reduced fertility potential, and about providing a semen sample for semen analysis. Semen analysis is the gold standard for fertility preservation in adult patients, but is only rarely considered by post-pubertal adolescent and young adult patients and their families. Only the semen analysis parameters will be used by the study for the comparison with physical and endocrine measures to assess whether spermatogenesis in these patients coincides with pubertal development. All potential frozen samples will be stored for the patient's future use, and samples will not be used for research experiments.

SUMMARY:
Klinefelter syndrome is characterized by primary testicular failure and progressive infertility. The objective of this study is to determine if sperm are present and can be observed in semen samples of adolescent and young adult Klinefelter patients and to determine whether the presence of sperm correlates with physical and/or clinically obtained hormone measures of pubertal development.

This study was designed in order to answer the following questions:

1. Is it possible to retrieve sperm for cryopreservation from semen samples of adolescent and young adult Klinefelter patients?
2. Does the presence of sperm correlate with the physical and/or endocrine measures that are assessed during routine clinical evaluations of pubertal development in the KS patient population?
3. If sperm retrieval is possible, what is the optimal age at which sperm retrieval should be attempted?

DETAILED DESCRIPTION:
Klinefelter Syndrome (KS) is a genetic condition in boys and men that results from having two X chromosomes and one Y chromosome. The incidence of the 47, XXY karyotype that defines the disorder ranges from 1:500 to 1:1000 in newborn males. The sexual development and fertility phenotypes of Klinefelter's syndrome include azoospermia (absence of sperm in the ejaculate), small firm testes, gynaecomastia (enlargement of breast tissue), low testosterone levels, and elevated follicle-stimulating hormone (FSH) and luteinizing hormone (LH) levels that can have an important impact on the quality of life for these patients. Beginning with puberty, testicular biopsies from Klinefelter patients progressively show a degenerated testicular environment with Sertoli-cell-only tubules, sclerotic or hyalinized tubules, and interstitial Leydig cell hyperplasia. Nevertheless, scattered areas with focal spermatogenesis can be seen in Klinefelter men, and assisted reproductive techniques now offer hope for patients who wish to father their own biological children. In these cases, a surgical sperm recovery procedure called testicular sperm extraction (TESE) is performed to extract sperm for in vitro reproductive methods. Success rates for testicular sperm extraction in Klinefelter patients are consistently above 50% (50 - 72%) and are similar to the success rates reported for TESE in azoospermic patients without Klinefelter syndrome. Pregnancy rates and life births after intracytoplasmic sperm injection (ICSI) are similar in couples with or without KS, and babies fathered by KS patients have a normal karyotype. Previous studies in adult KS patients reported that sperm recovery rates were significantly lower after the age of 35. Therefore, it was suggested that surgical sperm recovery in younger (possibly pubertal) boys should be considered as an option to maximize the opportunity to preserve their fertility before becoming sterile. However, there is considerable debate about the benefit of early invasive fertility intervention for KS patients.

The standard, non-invasive and safe way to obtain and analyze sperm production and quality in normal post-pubertal males is to obtain a semen sample by masturbation. It is currently unknown when spermatogenesis starts in boys with KS, and if sperm could be detected by semen analysis in early puberty. In this proposal, the investigators aim to determine if non-invasive methods during puberty could be useful to assess the reproductive potential of KS patients, and to possibly cryopreserve sperm from these patients for future use with well-established assisted reproductive techniques like in vitro fertilization with ICSI (intra cytoplasmic sperm injection).

Although this will be a sensitive topic for adolescent patients with KS and their parents, it is essential to begin the conversation regarding fertility preservation. Indeed, most parents and patients have questions regarding future fertility. This study has a secondary benefit in that it provides an ideal opportunity to educate the affected males and their families about the long-term effects of KS on their fertility and the availability of reproductive technologies to help with fertility. Similar discussions are becoming increasingly common (standard of care) for cancer patients who are at risk for infertility due to their disease or oncologic treatment.

It is currently unknown when spermatogenesis starts in boys with KS. While it seems to be commonly accepted that there is a progressive depletion of germ cells in the testes of KS patients after the onset of puberty, the data to support this notion are equivocal due to small patient populations, lack of controls and absence of longitudinal data.

In addition, the standard therapy for boys with KS is testosterone replacement therapy to trigger entry and progression of puberty characterized by the development of secondary sexual characteristics, bone maturation, and continued linear growth. However, testosterone supplementation also suppresses spermatogenesis (if present) through negative feedback on the hypothalamus-pituitary-gonadal axis. Some argue that any intervention to preserve fertility for KS patients should ideally precede hormone replacement therapy. However, in one study it was proposed that topical testosterone therapy might not negatively affect spermatogenesis in adolescent KS patients. The risks and unknowns of invasive surgical procedures like TESE for boys have to be carefully weighed against the possible benefits for this unique patient population. For these reasons, the investigators propose that non-invasive methods would be appropriate to retrieve sperm and are essential to gain insights about the initiation and decline of spermatogenesis in KS patients.

In this study, the investigators will analyse if sperm can be found in semen of Klinefelter patients during puberty and early adulthood. Participants will be followed until they reach age 26. During the time of their study participation, participants will provide at least one semen sample.

ELIGIBILITY:
Inclusion Criteria:

* males between the ages of 12 and 25
* diagnosed with mosaic or non-mosaic Klinefelter's Syndrome
* having bilaterally descended testes
* not having had a febrile illness within 3 months of enrollment.

Exclusion Criteria:

* previous treated with gonadotoxic chemotherapeutic or radiation regimen.
* psychological, psychiatric, or other conditions which prevent giving fully informed consent.

Ages: 12 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescent and young adults males who are proven to have Klinefelter Syndrome based on prior chromosome analysis (47,XYY).
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Presence of sperm in semen. | On average once a year until the participant turns 26
  Participants will provide at least one semen sample. The presence of sperm will be analyzed.
  Participants will also be given the opportunity to have their semen analysed for the presence of sperm once a year.
  Participants will be followed until they reach age 26.

SECONDARY OUTCOMES:
Longitudinal correlation of developmental and endocrine parameters with the presence or absence of sperm in semen samples. | 1 time a year for an average of 7.4 years
  Participants will be followed until they reach age 26. Thereafter, patients will be contacted once a year via phone to asses fertility/infertility issues and over all health.
Correlation of developmental parameters with the presence or absence of sperm in semen samples. | 1-2 times a year for an average of 7.4 years
  Participants will be scheduled for a routine visit with the endocrinologist 1-2 times a year.
  At each visit, the endocrinologist will measure height.
Correlation of developmental parameters with the presence or absence of sperm in semen samples. | 1-2 times a year for an average of 7.4 years
  Participants will be scheduled for a routine visit with the endocrinologist 1-2 times a year.
  At each visit, the endocrinologist will measure weight.
Correlation of developmental parameters with the presence or absence of sperm in semen samples. | 1-2 times a year for an average of 7.4 years
  Participants will be scheduled for a routine visit with the endocrinologist 1-2 times a year.
  At each visit, the endocrinologist will measure body proportions.
Correlation of developmental parameters with the presence or absence of sperm in semen samples. | 1-2 times a year for an average of 7.4 years
  Participants will be scheduled for a routine visit with the endocrinologist 1-2 times a year.
  At each visit, the endocrinologist will measure Tanner stages.
Correlation of developmental parameters with the presence or absence of sperm in semen samples. | 1-2 times a year for an average of 7.4 years
  Participants will be scheduled for a routine visit with the endocrinologist 1-2 times a year.
  At each visit, the endocrinologist will examine the presence of gynecomastia.
Correlation of developmental parameters with the presence or absence of sperm in semen samples. | 1-2 times a year for an average of 7.4 years
  Participants will be scheduled for a routine visit with the endocrinologist 1-2 times a year.
  At each visit, the endocrinologist will measure and bilateral testicular size.
Correlation of endocrine parameters with the presence or absence of sperm in semen samples. | 1-2 times a year for an average of 7.4 years
  Participants will be scheduled for a routine visit with the endocrinologist 1-2 times a year.
  At each visit, the endocrinologist will measure testosterone (T).
Correlation of endocrine parameters with the presence or absence of sperm in semen samples. | 1-2 times a year for an average of 7.4 years
  Participants will be scheduled for a routine visit with the endocrinologist 1-2 times a year.
  At each visit, the endocrinologist will measure luteinizing hormone (LH)
Correlation of endocrine parameters with the presence or absence of sperm in semen samples. | 1-2 times a year for an average of 7.4 years
  Participants will be scheduled for a routine visit with the endocrinologist 1-2 times a year.
  At each visit, the endocrinologist will measure follicle-stimulating hormone (FSH).
Correlation of endocrine parameters with the presence or absence of sperm in semen samples. | 1-2 times a year for an average of 7.4 years
  Participants will be scheduled for a routine visit with the endocrinologist 1-2 times a year.
  At each visit, the endocrinologist will measure serum anti-Mullerian hormone (AMH).
Correlation of endocrine parameters with the presence or absence of sperm in semen samples. | 1-2 times a year for an average of 7.4 years
  Participants will be scheduled for a routine visit with the endocrinologist 1-2 times a year.
  At each visit, the endocrinologist will measure inhibin B.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Orwig, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania